CLINICAL TRIAL: NCT03805334
Title: The Effectiveness of Bilateral Alternating Tactile Stimulation for Improving Sleep in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20013034
Record Dates: First submitted 2018-12-19; First posted 2019-01-15 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Sleep; Sensory Disorders
Keywords: sleep; sensory over-responsiveness; hypersensitivity
MeSH Terms: conditions — Sensation Disorders; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This study will use a non-concurrent multiple baseline design (MBD) where subjects will serve as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Touchpoints (Experimental): Subjects will wear Touchpoints devices on both ankles daily for 10 days. The devices will be worn ~1 hour before bedtime and through the night. They will be removed upon waking in the morning.
  Interventions: Other: Touchpoints

INTERVENTIONS:
Other: Touchpoints — Touchpoints are worn on either the wrists or ankles. They deliver a low level vibration in an alternating fashion to the skin.

SUMMARY:
The investigators hypothesize that wearing bilateral therapeutic vibrating devices before bed will result in positive changes in outcome measures related to sleep (e.g., sleep efficiency) in children who are sensitive to stimuli in their environment (aka sensory over responsiveness or SOR).

DETAILED DESCRIPTION:
The purpose of this research study is determine if providing bilateral alternating stimulation to the extremities is effective for improving sleep in children with sensory processing difficulties. The investigators will use Touchpoints to deliver the intervention. The Touchpoints look like a regular watch, and vibrate at different low level frequencies to produce a calming effect on the body. More information about Touchpoints can be found here: https://thetouchpointsolution.com/pages/shop-touchpoints. The investigators hypothesize that these types of wearable vibrating devices may help children fall asleep faster and possibly stay asleep longer. This study will allow the research team to test these assumptions.

In this study, each child will be asked to do the following things:

1. Wear an activity tracker watch on their wrist before bed and through the night for 10 days consecutively (Baseline)
2. Wear both the activity tracker watch (wrist) and the Touchpoints (both ankles) before bed and during sleep for 10 days straight. (Intervention)
3. Wear the activity tracker watch on their wrist before bed and through the night for 10 additional days (post-test)

During the study, the parents will be asked to fill out a brief sleep diary.

ELIGIBILITY:
Inclusion Criteria:

* Scores "more than others" in either sensation avoiding or sensory over-responsive on the Short Sensory Profile
* Has identified sleep difficulties on the Children's Sleep Wake Scale (any sub-scale scores outside of normative range)

Exclusion Criteria:

* Diagnosed seizure disorder or history of seizures
* Rubber or latex allergy (will not be able to wear wrist band)
* Significant motor impairments (e.g. cerebral palsy)
* Children who are wards of the state

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Short Sensory Profile 2 | Change from baseline to study completion (~30 days)
  The Short Sensory Profile 2 is a caregiver questionnaire for children ages 3-14 years. It draws questions from the Child Sensory Profile 2 which measures sensory processing on two intersecting scales: high vs. low threshold for responding to sensations and passive vs. active self-regulation in anticipation or response to sensory stimuli. The Short Sensory Profile 2 is primarily used for research and screening purposes while the Child Sensory Profile 2 is for clinical practice. The investigators will use this during the screening phase of the study to determine whether potential participants have sensory processing differences.
The Children's Sleep Wake Scale (CSWS) | Change from baseline to study completion (~30 days)
  The Children's Sleep-Wake Scale is a caregiver questionnaire for children ages 2-8 years. It covers children's going to bed, falling asleep, arousing and awakening during the night, returning to sleep after awakening during the night, and waking during the morning. The investigators will use this during the screening phase of the study to determine whether potential participants have trouble with sleep behaviors and to assess whether the intervention significantly changed sleep behaviors. The Children's Sleep Wake Scale includes a total of 25 questions that are ranked on a scale of 1 (never) to 6 (always). Five sub-scale scores are derived from this measure (Going to Bed, Falling Asleep, Maintaining Sleep, Re-initiating Sleep, Returning to Wakefulness) as well as a Total Sleep Quality score (mean of all 5 sub-scale scores added together). Both the sub-scales and the total scores are "reverse scored" (e.g., 1=6 and 6=1) so that higher scores equal better sleep quality.
Sleep Efficiency | Change from baseline to study completion (~30 days)
  Sleep efficiency is the ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed. Sleep efficiency will be measuring using the ActiGraph GT9X Link, a device that is worn like a watch that measures a person's activity. Efficiency will be reported as a percentage (e.g., 88% sleep efficiency). Scores above 85% are general considered within normal range; however each subject will serve as their own control and improvements will be noted from baseline to post-intervention.
Sleep Latency | Change from baseline to study completion (~30 days)
  Sleep latency refers to the time (measured in minutes) that it takes for a subject to fall asleep once they have "gone to bed". Sleep latency will be determined by comparing data that is recorded by the ActiGraph GT9X Link device (activity tracker) with data recorded by parents in the child's Sleep Diary. In the diary, parents will be asked to answer the following question: What time did you (or your child) try to go to sleep? This is usually when you turn the lights out and any devices off. Changes in sleep latency will be compared between baseline and intervention phases as well as at the completion of a post-intervention phase.
Number of Nighttime Awakenings | Change from baseline to study completion (~30 days)
  This is a count variable which will automatically be calculated by the ActiGraph GT9X Link device worn on the child's wrist. The ActiGraph will be programed to count any active movement lasting longer than 10 seconds after sleep has been initiated as a "nighttime awakening". Total number of night time awakenings will be compared across baseline, intervention, and post-intervention phases.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Reynolds, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Katherine Lawrence Dragas Sensory Processing and Stress Evaluation Lab, Richmond, Virginia, United States